CLINICAL TRIAL: NCT04408287
Title: Improving Activity Engagement Among Persons With SCI During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115929
Record Dates: First submitted 2020-05-20; First posted 2020-05-29 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; spinal cord injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: The proposed study will deliver an online physical activity program to persons with SCI across Ontario through the WebEx platform at Parkwood Institute. Participants will be recruited from across Ontario through SCI rehabilitation centers and established service providers. Strategic advertising through community partners such as Spinal Cord Injury Ontario, Canadian SCI Alliance and Ontario Neurotrauma Foundation will also be conducted. Study participants will include those with a spinal cord injury that have completed rehabilitation and are living in the community. Participants must have some upper limb function permitting arm movement against gravity. All participants must have physician clearance to participate in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The program will be delivered twice-weekly through 45-minute sessions over 6 weeks. An experienced fitness instructor with lived experience and a graduate student from the Department of Health and Rehabilitation Sciences, will lead a class of 4-6 participants. The sessions will be comprised of a 10-minute warm-up phase, a 25-minute aerobic phase and a 10-minute cool-down phase that will incorporate upper-extremity flexibility exercises and mindfulness meditation. Over the duration the instructor will be sensitive to varying levels of function and fitness and will structure the classes to enable a slow progression of intensity. Individual semi-structured interviews will be completed over the WebEx platform to garner feedback and improve study programming for future implementation of a health care service at Parkwood Institute Outpatient Clinic.
  Interventions: Other: WebEx Physical Activity Program

INTERVENTIONS:
Other: WebEx Physical Activity Program — The program will be delivered twice-weekly through 45-minute sessions over 6 weeks. An experienced fitness instructor with lived experience and a graduate student from the Department of Health and Rehabilitation Sciences, will lead a class of 4-6 participants. The sessions will be comprised of a 10-minute warm-up phase, a 25-minute aerobic phase and a 10-minute cool-down phase that will incorporate upper-extremity flexibility exercises and mindfulness meditation. Over the duration the instructor will be sensitive to varying levels of function and fitness and will structure the classes to enable a slow progression of intensity. Individual semi-structured interviews will be completed over the WebEx platform to garner feedback and improve study programming for future implementation of a health care service at Parkwood Institute Outpatient Clinic.

SUMMARY:
During the current COVID-19 pandemic many spinal cord injury (SCI) rehabilitation services are limited to emergency management, leaving those living in the community without access to services. Unfortunately, this can lead to negative effects including increase in emotional distress, feelings of isolation, and decreased activity engagement. Due to their limited mobility and greater likelihood of respiratory illness it is imperative to provide alternative forms of activity engagement to reduce their risk for secondary complications. Physical activity has been demonstrate to have numerous benefits for individuals with SCI ranging from enhanced health through prevention of secondary complications to improved subjective well-being. The current study proposes to provide an online physical activity program through web-based videoconferencing to person with SCI to improve overall wellbeing and activity engagement. The program will consist of six weeks of twice-weekly, 45-minute sessions in which an experienced fitness instructor (i.e., wheelchair aerobics) with lived experience and a Kinesiology graduate student will lead online sessions. The sessions will be comprised of a 10-minute warm-up phase, a 25-minute aerobic phase and a 10-minute cool-down phase that will incorporate upper-extremity flexibility exercises and guided meditation. In all cases, remote (i.e., in-home) participant monitoring of physiological signals will be conducted by the instructor to ensure safety of participants. Once the program has been completed, participants will be asked to complete self-report questionnaires related to acceptability, feasibility, and limited effectiveness. Participants will also be asked to complete a brief semi-structured interview examining barriers and facilitators of the program. Participant feedback from the interviews will be used to further develop of the program to meet the needs of the population and develop sustainable approaches for access to care in the community setting through collaborations with community partners (SCI Ontario, National SCI Alliance, Ontario Neurotrauma Foundation). Ultimately, the proposed project aims to improve overall wellbeing and access to health care service for those with SCI during the COVID-19 quarantine.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years or older; living with a spinal cord injury; living in the community in Ontario; access to a computer and internet

Exclusion Criteria:

* Not cleared by a physician to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment Satisfaction | 6 weeks
  Treatment Satisfaction Questionnaire

SECONDARY OUTCOMES:
Ability to Participate in Social Roles and Activities | Baseline, 6 weeks, and at 3 month follow-up
  Spinal Cord Injury - Quality of Life Short Form
Fatigue | Baseline, 6 weeks, and at 3 month follow-up
  Spinal Cord Injury - Quality of Life Short Form
Satisfaction with Social Roles and Activities | Baseline, 6 weeks, and at 3 month follow-up
  Spinal Cord Injury - Quality of Life Short Form
Positive Affect and Well-Being | Baseline, 6 weeks, and at 3 month follow-up
  Spinal Cord Injury - Quality of Life Short Form
Pain Interference | Baseline, 6 weeks, and at 3 month follow-up
  Spinal Cord Injury - Quality of Life Short Form
Resilience | Baseline, 6 weeks, and at 3 month follow-up
  Spinal Cord Injury - Quality of Life Short Form
Self-Esteem | Baseline, 6 weeks, and at 3 month follow-up
  Spinal Cord Injury - Quality of Life Short Form

OTHER OUTCOMES:
Fear of COVID-19 Scale | Baseline, 6 weeks, and at 3 month follow-up
  Fear of COVID-19 Scale

CONTACTS AND LOCATIONS:
Overall Officials: Swati Mehta, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Eldon Loh, PhD, Principal Investigator — Parkwood Institute, St. Joseph's Health Care London
Locations (1):
- St. Josephs Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No